CLINICAL TRIAL: NCT03473002
Title: A Phase I Double-Blind Placebo Controlled Trial to Evaluate the Safety and Immunogenicity of Intranasal Sendai Virus Vectored Respiratory Syncytial Virus (SeVRSV) Vaccine in Healthy Adults
Brief Title: A Safety and Immunogenicity Study of Intranasal Sendai Virus Vectored Respiratory Syncytial Virus (SeVRSV) Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-0108; HHSN272201300016I
Record Dates: First submitted 2018-03-15; First posted 2018-03-21 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-03-05

CONDITIONS: Antiviral Prophylaxis; Respiratory Syncytial Virus Infection
Keywords: Immunogenicity; Respiratory Syncytial Virus; Safety; Sendai Virus; Vaccine
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): One dose of placebo (0.9% Sodium Chloride) intranasally, n=4
  Interventions: Other: Placebo
- SeVRSV (Experimental): 1 x 10^7 EID50 (one dose) of SeVRSV vaccine intranasally, n=16
  Interventions: Biological: SeVRSV Vaccine

INTERVENTIONS:
Other: Placebo — 0.9% Sodium Chloride
  Arms: Placebo
Biological: SeVRSV Vaccine — Recombinant Sendai virus vectored respiratory syncytial virus (SeVRSV) vaccine. SeVRSV is a replication-competent Sendai virus that carries the RSV F gene produced by reverse genetics technology.
  Arms: SeVRSV

SUMMARY:
This is a Phase I randomized, double blind, placebo controlled trial in up to 25 males and non-pregnant females, 18-45 years old, inclusive, who are in good health and meet all eligibility criteria. This trial is designed to assess the safety, reactogenicity and immunogenicity of a single intranasal dose of Sendai virus vectored Respiratory Syncytial Virus (SeVRSV) vaccine. The subjects will be randomized in a 4:1 ratio to receive SeVRSV vaccine at a dose of 1 x 10^7 EID50 or placebo (saline) intranasally. Study duration is approximately 11 months with subject participation duration approximately 6 months. The primary objectives are to: 1) assess the safety and reactogenicity of SeVRSV vaccine following receipt of one intranasal dose; 2) assess the ELISA antibody responses to SeV and to the RSV F protein at 28 days post receipt of one intranasal dose of SeVRSV vaccine; 3) assess the detection of vaccine virus from nasal washes at days 3, 5, 8 and 15 following receipt of one intranasal dose of SeVRSV vaccine.

DETAILED DESCRIPTION:
This is a Phase I randomized, double blind, placebo controlled trial in up to 25 males and non-pregnant females, 18-45 years old, inclusive, who are in good health and meet all eligibility criteria. This trial is designed to assess the safety, reactogenicity and immunogenicity of a single intranasal dose of Sendai virus vectored Respiratory Syncytial Virus (SeVRSV) vaccine. The subjects will be randomly assigned in a 4:1 ratio to receive SeVRSV vaccine at a dose of 1 x 10^7 EID50 or placebo (saline) intranasally. Since this is a first in human, phase I study, the first two subjects (sentinels) will be enrolled in the SeVRSV treatment arm. Safety and laboratory data will be collected through 14 days post vaccination. If none of the predefined halting criteria of sentinel subjects are met, enrollment of the remaining subjects will proceed. If any of the pre-defined halting criteria of sentinel subjects are met, an electronic review by the SMC will be required prior to continuation of the study. While safety is evaluated for the sentinel subjects, no new subjects will be enrolled, but screening may continue. Study duration is approximately 11 months with subject participation duration approximately 6 months. The primary objectives are to: 1) assess the safety and reactogenicity of SeVRSV vaccine following receipt of one intranasal dose; 2) assess the ELISA antibody responses to SeV and to the RSV F protein at 28 days post receipt of one intranasal dose of SeVRSV vaccine; 3) assess the detection of vaccine virus from nasal washes at days 3, 5, 8 and 15 following receipt of one intranasal dose of SeVRSV vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before initiation of any study procedures. 2. Are able to understand and comply with planned study procedures and be available for all study visits/phone calls.

3. Males or non-pregnant females 18-45, inclusive. 4. Are in good health.

* As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days that would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days. This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (with the exception of steroids as outlined in the Subject Exclusion Criteria), herbals, vitamins, and supplements are permitted.

  5. Oral temperature is less than 100.0 degrees Fahrenheit. 6. Pulse is 47 to 105 beats per minute (bpm), inclusive. 7. Systolic blood pressure (BP) is 85 to 150 mm Hg, inclusive. 8. Diastolic blood pressure (BP) is 55 to 95 mmHg, inclusive. 9. Women of childbearing potential must use an acceptable method of contraception from 30 days prior to study vaccination until 60 days after study vaccination.
  * Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy, or successful Essure (R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or < 1 year of the last menses if menopausal.

    --- Includes, but is not limited to, non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with a vasectomized partner, male condoms with the use of applied spermicide, intrauterine devices, NuvaRing (R), and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").

    10. Female subjects of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to study vaccination.

    11. Sexually active males with a woman of childbearing potential and has not had a vasectomy performed > 1 year prior to screening must agree not to father a child for 60 days after vaccination.
    * See criteria of women of childbearing potential above. ----- Must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner uses occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.

      11. Erythrocyte sedimentation rate (ESR) is less than 30 mm per hour. 12. White blood cells (WBC) are greater than 4.4 x 10^3/uL and less than 11.1 x 10^3/uL.

      13. Hemoglobin (Hgb) is greater than 11.6 g/dL for females or is greater than 13.2 g/dL for males.

      14. Platelets are greater than 134 x 10^3/uL and less than 466 x 10^3/uL. 15. Absolute Neutrophil Count is greater than 1.7 x 10^3/uL

      ------ For subjects who are of African American or Middle Eastern decent, ANC must be greater than 0.8 x 10^3/uL for inclusion.

      16. Alanine aminotransferase (ALT) is less than 1.25 ULN for females and males. 17. Aspartate aminotransferase (AST) is less than 1.25 ULN for females and males.

      18. Total bilirubin is less than 1.11 mg/dL. 19. Creatinine is less than 0.96 mg/dL for females or is less than 1.18 mg/dL for males.

      20. Sodium is greater than 135 mmol/L and less than 146 mmol/L. 21. Potassium is greater than 3.4 mmol/L and less than 5.2 mmol/L. 22. BUN is less than 19 mg/dL (BUN will be obtained only if creatinine is above normal range).

      23. HgbA1C is less than 6.3%. 24. Have normal screening laboratories for urine protein. Trace protein is acceptable.

      25. Drug screen for opiates is negative. 26. Have a normal ECG.
      * Abnormal screening electrocardiogram (ECG) defined as pathologic Q waves and significant ST-T wave changes: criteria for left ventricular hypertrophy; and any non-sinus rhythm excluding isolated premature atrial contractions.

        27. Agrees not to participate in another clinical trial during the study period.

        28. Agrees not to donate blood or blood products to a blood bank for 6 months after receiving the vaccine.

Exclusion Criteria:

1. Have an acute illness, as determined by the site PI or appropriate sub-investigator, within 72 hours prior to study vaccination.

   - An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol. Subjects may re-screen after an acute illness is resolved.
2. Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation.

   -- Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study.
3. History of anatomic disorder of the nares or nasopharynx (Deviated septum is allowed).
4. History of chronic sinus infections.
5. A diagnosis of type I or II diabetes.
6. Have a body mass index (BMI) < 18.5 or > / = 35 kg/m^2.
7. History of medical diagnosis of selected respiratory diseases.

   --- Asthma as an adult (defined as diagnosis at > / = 18 years of age), reactive airway disease, wheezing requiring medication as an adult (defined as diagnosis at > / = 18 years of age), cystic fibrosis, bronchopulmonary dysplasia, chronic pulmonary disease, medically confirmed apnea, hospitalization for respiratory illness or mechanical ventilation for respiratory illness.
8. History of smoking in the last 5 years.
9. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
10. Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma skin cancers that are not active are permitted.
11. Positive hepatitis C, or HIV serology or positive hepatitis B serology not consistent with prior hepatitis B immunization.
12. History of Bell's Palsy.
13. History of anosmia (per subject report of ever having symptoms or clinician diagnosis).
14. Have known hypersensitivity or allergy to eggs, or other components of the study vaccine.
15. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
16. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
17. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
18. Have taken oral or parenteral (including intraarticular) corticosteroids of any dose within 30 days prior to study vaccination.
19. Have taken high-dose inhaled corticosteroids within 30 days prior to study vaccination.

    ---- High-dose defined using the inhaled high-dose reference chart.
20. Receipt of any intranasal medication within 7 days prior to study vaccination through 14 days post study vaccination.
21. Received any licensed live vaccine within 30 days of study vaccination.
22. Received a licensed inactivated vaccine within 14 days of the study vaccination.
23. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to study vaccination.
24. Received an experimental agent within 28 days prior to study vaccination, or expects to receive an experimental agent during the 6-month trial-reporting period.

    ----- Including vaccine, drug, biologic, device, blood product, or medication.

    ------ Other than from participation in this study.
25. Female subjects who are breastfeeding or plan to breastfeed at any given time from the receipt of study vaccination throughout the 6 month trial period.
26. Expected household contact or same room contact for > 1 hour with children < 6 months of age or immunocompromised individuals within 7 days of receipt of study vaccination.
27. Day care provider or healthcare provider with direct contact with children or patients.
28. Have received any antiviral drug within 3 days of study vaccination.
29. Any condition that would, in the opinion of the Site Investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Occurrence of clinical safety laboratory abnormalities | Up to 7 days
Occurrence of Medically Significant Wheezing | Up to 6 months
Occurrence of New Onset Chronic Medical Conditions (NOCMCs) | Up to 6 months
Occurrence of SAEs not related to study product | Up to 6 months
Occurrence of solicited local reactogenicity | Up to 14 days
Occurrence of solicited systemic reactogenicity | Up to 14 days
Occurrence of unsolicited adverse events | Up to day 28
Occurrence of vaccine-related SAEs | Up to 6 months
Percentage of subjects achieving a 4 - fold rise in RSV F antibody titer measured by ELISA | From day 1 through day 29
Percentage of subjects achieving a 4 - fold rise in SeV antibody titer measured by ELISA | From day 1 through day 29
Percentage of subjects with vaccine virus detected by nasal wash assessed by Polymerase Chain Reaction (PCR) | Day 15
Percentage of subjects with vaccine virus detected by nasal wash assessed by Polymerase Chain Reaction (PCR) | Day 3
Percentage of subjects with vaccine virus detected by nasal wash assessed by Polymerase Chain Reaction (PCR) | Day 5
Percentage of subjects with vaccine virus detected by nasal wash assessed by Polymerase Chain Reaction (PCR) | Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio, United States